CLINICAL TRIAL: NCT00489060
Title: A Randomized Trial of External Beam Radiotherapy Versus Cryoablation in Patients With Clinically Localized Prostate Cancer
Brief Title: A Randomized Trial of External Beam Radiotherapy Versus Cryoablation in Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Cancer Trials Group (Network); AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9716
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2008-07-17 (Estimated); Status verified 2008-07

CONDITIONS: Prostate Cancer
Keywords: Cryoablation; Radiation; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Cryoablation and External Beam Radiation

SUMMARY:
A trial to determine if cryoablation is as effective as radiation in the treatment of men with localized prostate cancer.

DETAILED DESCRIPTION:
Men with newly diagnosed localized prostate cancer were randomly assigned to cryoablation or external beam radiotherapy (median dose 68 Gy). All patients received neoadjuvant antiandrogen therapy. The primary endpoint was disease progression at 36 months based on a trifecta definition of failure: (a) radiological evidence of metastatic disease or b) initiation of further antineoplastic therapy or c) biochemical failure). Two definitions of biochemical failure were used: 1) rising PSA with a final value >1.0 ng/mL and 2) rise above PSA nadir + 2 ng/mL. Secondary endpoints were overall survival, disease-specific survival, and positive prostate biopsy at 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinically localized prostate cancer
* PSA < 20ng/ml
* Negative bone scan

Exclusion Criteria:

* Previous TURP
* Previous hormone therapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 1997-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
No evidence of disease progression (NEDP) at 36 months | 36 months

SECONDARY OUTCOMES:
Prostate biopsy status | 36 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Donnelly, MD, Principal Investigator — Tom Baker Cancer Center
Locations (1):
- Tom Baker Cancer Center, Calgary, Alberta, Canada